CLINICAL TRIAL: NCT00108823
Title: A 24-week, Double Blind, Randomized Study to Investigate the Effect of 500 µg Roflumilast Tablets Once Daily Versus Placebo on Parameters Indicative of Hyperinflation in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: The HERO-study: Effects of Roflumilast in Patients With COPD (Chronic Obstructive Pulmonary Disease) (BY217/M2-121)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-121
Record Dates: First submitted 2005-04-19; First posted 2005-04-20 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

INTERVENTIONS:
Drug: Roflumilast

SUMMARY:
The purpose of this trial is to study the effects of roflumilast on lung function parameters indicative of hyperinflation in patients with COPD.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* Patients with a history of chronic obstructive pulmonary disease for at least 12 months as defined by the GOLD (Global Initiative on Obstructive Lung Diseases) criteria (2003)
* Age ≥ 40 years
* FEV1/FVC ratio (post-bronchodilator) ≤ 70%
* FEV1 (post-bronchodilator) ≤ 65% of predicted
* FRC (post-bronchodilator) ≤ 120% of predicted
* Clinically stable COPD within 4 weeks prior to baseline visit (B0).
* Availability of a chest x-ray dated a maximum of 6 months prior to study baseline visit (B0) or a willingness to have a chest x-ray performed at visit (B0).

Main Exclusion Criteria:

* COPD exacerbation indicated by a treatment with systemic glucocorticosteroids not stopped at least 4 weeks prior to the baseline visit (B0)
* Non smoker, current smoker or ex-smoker (smoking cessation at least one year ago) with a smoking history of < 10 pack years
* Suffering from any concomitant disease that might interfere with study procedures or evaluation
* Lower respiratory tract infection not resolved 4 weeks prior to the baseline visit (B0)
* Diagnosis of asthma and/or other relevant lung disease (e.g. history of bronchiectasis, cystic fibrosis, bronchiolitis, lung resection, lung cancer, interstitial lung disease [e.g. fibrosis, silicosis, sarcoidosis], and active tuberculosis)
* Current participation in a pulmonary rehabilitation program or completion of a pulmonary rehabilitation program within 2 months preceding the baseline visit (B0).
* Known alpha-1-antitrypsin deficiency
* Need for long term oxygen therapy defined as ≥ 15 hours/day
* Clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical evaluation (as assessed by the investigator)
* Known infection with HIV, active hepatitis and/or liver insufficiency
* Diagnosis or history of cancer (other than basal cell carcinoma) or recurrence within 5 years prior to study start
* Clinically significant cardiopulmonary abnormalities (diagnosed clinically or by x-ray/ECG) that are not related to COPD and that require further evaluation
* Pregnancy, breast feeding, oocyte donation or oocyte implantation planned during the trial
* The female patient is of childbearing potential and is not using and is not willing to continue to use a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, unless she is surgically sterilized/hysterectomized or post-menopausal > 1 year or any other criteria considered sufficiently reliable by the investigator in individual cases
* Participation in another study (use of investigational product) within 30 days preceding the baseline visit (B0) or re-entry of patients already enrolled in this trial
* Suspected inability or unwillingness to comply with study procedures
* Alcohol or drug abuse
* Inability to follow study procedures due to, for example, language problems or psychological disorders
* Use of prohibited drugs
* Suspected hypersensitivity to the study medication and/or contraindication to any ingredients of the study medication (roflumilast) or rescue medication

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550
Dates: Start 2004-10

PRIMARY OUTCOMES:
Lung function parameters indicative of hyperinflation in patients with COPD

SECONDARY OUTCOMES:
Mean change from randomization to endpoint in additional pre and post bronchodilator spirometric and lung volume parameters
Measurement of quality of life parameters and dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (16):
- United States (10):
  - ALTANA Pharma, Cities in California, California
  - ALTANA Pharma, Cities in Colorado, Colorado
  - ALTANA Pharma, Cities in Florida, Florida
  - ALTANA Pharma, Cities in Missouri, Missouri
  - ALTANA Pharma, Cities in New Mexico, New Mexico
  - ALTANA Pharma, Cities in New York, New York
  - ALTANA Pharma, Cities in Oregeon, Oregon
  - ALTANA Pharma, Cities in South Carolina, South Carolina
  - ALTANA Pharma, Cities in Texas, Texas
  - ALTANA Pharma, Cities in Washington, Washington
- ALTANA Pharma, Cities in Canada, Canada
- ALTANA Pharma, Cities in France, France
- ALTANA Pharma, Cities in Poland, Poland
- ALTANA Pharma, Cities in South Africa, South Africa
- ALTANA Pharma, Cities in Spain, Spain
- ALTANA Pharma, Cities in the United Kingdom, United Kingdom

REFERENCES:
- See also: BY217-M2-121-RDS-2008-12-23.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4479&filename=BY217-M2-121-RDS-2008-12-23.pdf